CLINICAL TRIAL: NCT02020590
Title: A Pilot Phase 1/2a, Multicentre, Open Proof-of-concept Study on the Efficacy and Safety of Allogeneic Osteoblastic Cells (ALLOB®) Implantation in Non-infected Delayed-Union Fractures
Brief Title: Phase 1/2a Study on Allogeneic Osteoblastic Cells Implantation in Delayed-Union Fractures
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bone Therapeutics S.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLOB-DU1
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Results first posted 2021-09-28 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Long Bone Delayed-Union Fracture
Keywords: Delayed-Union Fractures; Impaired Healing; Fractures; Orthopedics; Bone; Musculoskeletal Disorders
MeSH Terms: conditions — Fractures, Bone; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALLOB® Implantation (Experimental): One arm: ALLOB® Implantation
  Interventions: Drug: ALLOB® implantation

INTERVENTIONS:
Drug: ALLOB® implantation — Each patient will undergo a single administration of ALLOB® into the delayed-union site under anesthesia.

SUMMARY:
Fracture healing is a complex physiological process caused by interaction of cellular elements, cytokines and signaling proteins, which results in the formation of new bone. There is for now no universally accepted approach to evaluate the progression of fracture healing. Typically, a fracture is considered as a delayed-union when the bone has not united within a period of time that would be considered adequate for bone healing. Delayed-union suggests that union is slow but will eventually occur without additional surgical or non-surgical intervention, whereas non-union is defined as the cessation of all reparative process of healing.

The incidence of impaired healing is estimated to range from 5 to 10% of all long bone fractures, depending on the fracture site, the type and degree of injury, among other factors. Currently the treatment of choice remains bone allograft or autograft. This procedure shows in general good results but requires an invasive surgery of several hours under general anesthesia, followed by a few days of hospitalization. Because of this, major complications have been reported in up to 20-30% of patients.

The present Phase 1/2a study aims at demonstrating the safety and efficacy of ALLOB®, a proprietary population of allogeneic osteoblastic cells, in the treatment of delayed-union fractures of long bones. In this study, delayed-union is defined at the time of screening as an absence of healing of minimum 3 months and maximum 7 months (+/- 2 weeks) after the onset of the fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patient (or patient's legally acceptable representative) capable to provide a written, dated, and signed informed consent prior to any study related procedure
* Non-infected delayed-union fracture of a long bone of minimum 3 months and maximum 7 months (+/- 2 weeks)

Exclusion Criteria:

* Fracture interline larger than 2.5 cm
* Insufficient fracture stability
* Multifocal fracture
* Positive serology for hepatitis B, hepatitis C, Human Immunodeficiency Virus (HIV)
* Current or past medical disease that could interfere with the evaluation of the safety and efficacy, as judged by the investigator
* Severe renal or hepatic impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02; Primary Completion 2017-09 (Actual); Study Completion 2020-01-30 (Actual)

REFERENCES:
- [Derived] Jayankura M, Schulz AP, Delahaut O, Witvrouw R, Seefried L, Berg BV, Heynen G, Sonnet W. Percutaneous administration of allogeneic bone-forming cells for the treatment of delayed unions of fractures: a pilot study. Stem Cell Res Ther. 2021 Jun 26;12(1):363. doi: 10.1186/s13287-021-02432-4. PMID 34174963

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 25 patients enrolled in the study (ICF signature), 22 patients were treated:
  * 2 patients were considered as non eligible before treatment
  * 1 patient withdrew consent before prior to Day 0
Period: Overall Study
Arm/Group | ALLOB® Implantation
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population (all patients treated)
Arm/Group | ALLOB® Implantation
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (13.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 22
Region of Enrollment [Number; unit: participants]
  Belgium | 13
  Germany | 9
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.73 (4.676)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders at 6 Months (Efficacy of ALLOB)
Description: The success of the study will be based on the percentage of treated patients (ALLOB®) not failing under treatment. A patient will be considered as failed under treatment if, at Month 6: - He/she had a rescue surgery Or - The Global Disease Evaluation score (VAS) as perceived by the patient has not improved by at least 25% and the Tomographic Union Score (TUS) as assessed by CT scan has not increased by at least two points (versus baseline).
Time Frame: 6 months
Population: The efficacy analysis was conducted on the Per Protocol population (21 treated patients; one patient being excluded from the analysis due on a major protocol deviation)
Measure: Number (90% Confidence Interval); unit: percent of patients
Arm/Group | ALLOB® Implantation
Number analyzed (Participants) | 21
percent of patients | 100 [86.71 to 100]
Statistical Analysis 1: Comparison: ALLOB® Implantation; The success of ALLOB® treatment was based on the percentage of responders. A treated patient was considered as responding if, at the end of the study (6 months): * He/she had not required rescue surgery and * The GDE score as perceived by the patient had improved by at least 25% or the TUS (tomographic union score) as assessed by CT scan had increased by at least 2 points; Test type: Other; The response rate at Month 6 for the 21 patients in the PP population was 100 % (CI: 86.71 - 100.0%). None of the treated patients required rescue surgery. An improvement of GDE score of at least 25% was reported for 16 (76.2%) patients. An increase in TUS of at least 2 points was reported for 16 (76.2%) patients; all patients met at least one of these two criteria

ADVERSE EVENTS:
Time Frame: 6 months
Description: Emergence was defined from the date of ALLOB® implantation up to end of study visit (Month-6 visit)
Arm/Group | ALLOB® Implantation
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 2/22
Other Adverse Events (participants affected / at risk) | 9/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALLOB® Implantation (N=22)
implant site infection (Infections and infestations) | 1 (1)
angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALLOB® Implantation (N=22)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT02020590/Prot_SAP_000.pdf